CLINICAL TRIAL: NCT00690651
Title: Randomized Controlled Study Into Early Mobilization Following Internal Fixation of Isolated Ankle Fractures.
Brief Title: Rest Easy: Is Bed Rest Really Necessary After Surgical Repair of an Ankle Fracture?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Alfred (Other)
Collaborators: National Trauma Research Institute (Other)
Responsible Party: Ms Lara kimmel, The Alfred
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 166/08
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-01

CONDITIONS: Ankle Injuries; Fracture
Keywords: ankle; fracture; mobilisation; bed rest; internal fixation
MeSH Terms: conditions — Ankle Injuries; Fractures, Bone | interventions — Early Ambulation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): this group will rest in bed with operated leg well elevated for 48 hour and then mobilize with physiotherapist with aim for discharge home when safe.
  Interventions: Procedure: Standard mobilization
- 1 (Experimental): mobilize with physiotherapist within 24 hours of surgical fixation of fractured ankle
  Interventions: Procedure: Early mobilization

INTERVENTIONS:
Procedure: Early mobilization — pt to get out of bed and mobilize with physiotherapist within 24 hours of surgery. they will be allowed toilet privileges and will go home when safe (as per medical staff and allied health)
  Arms: 1
Procedure: Standard mobilization — this group will rest in bed with their leg elevated above their heart for 48 hours post surgery to ankle fracture and will then mobilize with physiotherapist with aim to discharge home.
  Arms: 2

SUMMARY:
After a patient has fractured an ankle that then requires surgery, the recommendation is to remain in bed, with the operated leg elevated on pillows for 48 hours. This is a precautionary measure, as yet unsubstantiated by research, which is thought to minimize ankle swelling that can inhibit the healing of the surgical wound. However, prolonged bed rest can lead to other complications such as blood clots in the lungs or leg veins, or chest infections such as pneumonia. Prolonged bed rest is also known to cause weakness and a loss of fitness such that recovery may be slower. In this research the investigators will be randomly allocating patients to mobilize within 24 hours post operatively or to rest in bed for 48 hours with their leg well elevated. The investigators will measure length of stay and wound healing and integrity at 14 days. This study aims to investigate whether getting patients out of bed within 24 hours of surgery can accelerate recovery and reduce acute hospital length of stay without affecting wound healing. If bed rest for 2 days is not necessary, there will be benefits for the patient in terms of general health and ability, and for the hospital in terms of cost savings through shorter lengths of stay and patient through put. The investigators already know that early mobilization is beneficial following other types of orthopedic surgery such as hip fractures. This study aims to investigate if early mobilization following surgical management of ankle fractures is safe with specific regard to wound integrity and wound outcomes. This study will also investigate the effect of earlier mobilization on the length of time spent in the acute hospital and for those discharged directly home, the amount and type of support required. If early mobilization is found to be safe for wound healing and results in shorter in-hospital stays, this research will provide the confidence to endorse a change to current clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* patients who have had internal fixation of a fractured ankle closed without plastic surgery intervention and without follow up hyperbaric oxygen therapy

Exclusion Criteria:

* living in nursing home,
* previously non-ambulant,
* concommitant injuries which do not allow early mobilisation, plastics involvement for wound closure, hyperbaric oxygen therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
length of acute hospital stay | various
  The time frame is variable as the length of stay is variable depending on many factors (usually less than a week in acute hospital if no complications)

SECONDARY OUTCOMES:
wound integrity | 10-14 days
readmission rate | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Lara a Kmmel, BA. Physio, Principal Investigator — Bayside Health; Anne Holland, Dr Physio, Study Director — Bayside Health
Locations (1):
- The Alfred, Melbourne, Victoria, Australia